CLINICAL TRIAL: NCT06585254
Title: Use of Transcutaneous Vagus Nerve Stimulation in Reducing the Symptoms of Long COVID Patients Who Fulfill Diagnostic Criteria for ME/CFS
Brief Title: tVNS in Long COVID-19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Benjamin Natelson, Professor of Neurology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY-23-01007
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-04

CONDITIONS: Long COVID; Chronic Fatigue Syndrome
Keywords: Medically unexplained illness; Vagus Nerve
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue Syndrome, Chronic

STUDY DESIGN:
Intervention Model Description: Randomized 6-week trial of two stimulus parameters in improving the health of PASC patients with CFS. Based on participation, then an additional 6 weeks using the device that had the best outcome in improving the health of PASC patients with CFS.
Who Masked: Participant, Outcomes Assessor
Masking Description: A computer-generated randomization list will be used to assign subjects into Treatment A or Treatment B. Study team members doing outcome assessments will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- #1: Patient controlled (Experimental): Patient will ramp up current intensity until uncomfortable, then ratchet back to what is comfortable and press button. Patient is to do this daily for 35 minutes for 6 weeks.
  Interventions: Device: Transcutaneous vagus nerve stimulator
- #2: Device Controlled (Experimental): Patients will ramp up current intensity until uncomfortable, then ratchet back to what is comfortable and press button. The device has software embedded in it that is used to arrive at a personalized way of stimulating the vagus nerve. At this level, the device stimulus will not be sensed by the patient. Patient is to do this daily for 35 minutes for 6 weeks.
  Interventions: Device: Transcutaneous vagus nerve stimulator

INTERVENTIONS:
Device: Transcutaneous vagus nerve stimulator — A device attached to the tragus of the ear which when activated stimulates an ascending branch of the vagus nerve

SUMMARY:
A prior open label study has shown that transcutaneous vagus nerve stimulation [tVNS] can improve the health of some patients with postacute sequelae of SARS-CoV-2 infection (PASC), severely affected enough to also fulfill criteria for myalgic encephalomyelitis / chronic fatigue syndrome (ME/CFS). The purpose of this study is to compare two sets of stimulus parameters to determine the one that best improves the health-related quality of life of these patients over a period of 6-weeks. Patients using their assigned device for at least 30 of the 42 possible opportunities will receive the best device for an additional 6-week period.

DETAILED DESCRIPTION:
While the US has officially said the SARS CoV-2 emergency is over, the country is left with a residual of patients who continue to experience Post-Acute Sequelae of SARS CoV-2 infection -- PASC. Unfortunately, despite a major effort to understand PASC via the NIH Researching Covid to Enhance Recovery program, no specific treatment has emerged and only a limited number of new trials has been initiated. The purpose of this proposal is to perform a clinical trial of noninvasive, transcutaneous vagus nerve stimulation [tVNS] in an attempt to find the best tVNS treatment for these patients.

The need for the proposed trial is supported by an earlier open label tVNS trial in 15 PASC patients who also fulfilled the 1994 case criteria for myalgic encephalomyelitis/chronic fatigue syndrome [ME/CFS but for simplicity CFS]. The research team chose patients with PASC-CFS for two reasons: first, CFS following Covid infection is probably the most common subgroup of patients with PASC. In the study, of 41 PASC patients whose continued symptoms over time lead to their being referred for cardiopulmonary exercise tests, 47% fulfilled the 1994 case criteria for the diagnosis of CFS. Second, the research team limited the tVNS pilot to PASC-CFS to reduce the heterogeneity inherent in the diagnosis of PASC. The research team specifically recruited non-hospitalized patients with documented Covid who remained ill with fatigue, widespread pain, cognitive complaints, and post-exertional malaise for at least 6 months after the acute infection, thus fulfilling the 1994 case criteria for CFS. Importantly, the entire study was done remotely without requiring participants to come into the medical center or stop current medical treatments.

The research team proposes to extend this study to inform us which of two possible ways of stimulating the vagus is the most effective in improving the health of PASC-CFS patients. The study again will be done remotely with the study team having access to large databases of non-hospitalized PASC sufferers. After determination that a patient had Covid, continued ill with PASC and now fulfills criteria for the diagnosis of CFS, the participant will be asked to respond to questionnaires via RedCap as to magnitude of fatigue, cognitive dysfunction, widespread pain and/or post-exertional malaise, as well as their functional status. Each will then be randomized into Treatment A or B and sent the device for these two treatment limbs with instructions to use the device for 35 min a day in the morning over a 6-week period.

During the fifth week of study participation, participants will receive a stick-on device [as well as instructions via zoom] to allow them to use the device to provide data on heart rate variability - an objective measure of treatment success. Participants will do this for a 6-minute period in the afternoon and then return the device to the study team.

Participants will complete questionnaires on RedCap at the end of the first 6-week phase and return the device to the study team to determine usage. Participants will be told they must use their device for at least 30 of the 42 days in order to get access to the device that gave the best clinical outcome for an additional 6-weeks. At the end of this second 6-week period, participants will again complete questionnaires and return their device to the study team.

ELIGIBILITY:
Inclusion Criteria:

* Must have had documented Covid infection and then fulfill 2015 case definition for ME/CFS
* Chalder Fatigue Scale score of 4 or greater
* SF-36 Physical Function scale score ≤70
* VAS values of 3 or higher from 0 [none] 3 [substantial] to 5 [very severe burden] on at least two of the following symptoms - fatigue; widespread pain, brain fog, post-exertional malaise

Exclusion Criteria:

* BMI ≥30
* Hospitalized for COVID-19 infection
* BMI ≥30
* Pregnancy

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The Chalder Fatigue Questionnaire (CFQ) | Baseline, at 6 week (end of blinded phase), and at 12 weeks (end of open label phase)
  The Chalder Fatigue Questionnaire (CFQ) is used as a measure of fatigue. The CFQ consists of 11 items and uses likert scoring 0, 1, 2, 3, providing a full scale range of 0-33, where lowest score is least fatigue.
Change in Short Form Health Survey (SF-36) | Baseline, at 6 week (end of blinded phase), and at 12 weeks (end of open label phase)
  The SF-36 is a multi-purpose, short form health survey consisting of 36 questions. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability. SF-36 will be assessed for physical function score improved from baseline by 0.6 SD or 14%.
Visual Analog Scale (VAS) measuring Fatigue | Baseline, at 6 week (end of blinded phase), and at 12 weeks (end of open label phase)
  VAS total scale from 0-5 scoring system [0 none; 1 mild; 2 moderate; 3 substantial; 4 severe; 5 very severe]. Higher score indicates poorer health outcome.
VAS to measure Widespread Pain | Baseline, at 6 week (end of blinded phase), and at 12 weeks (end of open label phase)
  VAS total scale from 0-5 scoring system [0 none; 1 mild; 2 moderate; 3 substantial; 4 severe; 5 very severe]. Higher score indicates poorer health outcome.
VAS measuring Postexertional malaise (PEM) | Baseline, at 6 week (end of blinded phase), and at 12 weeks (end of open label phase)
  VAS total scale from 0-5 scoring system [0 none; 1 mild; 2 moderate; 3 substantial; 4 severe; 5 very severe]. Higher score indicates poorer health outcome.
VAS measuring brain fog | Baseline, at 6 week (end of blinded phase), and at 12 weeks (end of open label phase)
  VAS total scale from 0-5 scoring system [0 none; 1 mild; 2 moderate; 3 substantial; 4 severe; 5 very severe]. Higher score indicates poorer health outcome.
Global Clinical Assessment of Change | At 6 week (end of blinded phase) and at 12 weeks (end of open label phase)
  Global Clinical Assessment of Change --+3 or +2 on a scale ranging from +3 [very much improved] thru 0 [no change] to -3 [very much worse]

SECONDARY OUTCOMES:
Heart Rate Variability (HRV) | Baseline and at 5-6 week (end of blinded phase)
  Participants will attach a device invented by the co-investigator which detects ECG and can quantify R-R intervals compute root mean square of successive differences (RMSSD) between normal heartbeats. The RMSSD reflects the beat-to-beat variance in heart rate and is the primary time-domain measure used to estimate the vagally mediated changes reflected in heart rate (HR).

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin H Natelson, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Anna Norweg, PhD, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  To achieve aims in the approved proposal. Proposals should be directed to anna.norweg@mssm.edu. To gain access, data requestors will need to sign a data access agreement.